CLINICAL TRIAL: NCT01469650
Title: Serum 25-hydroxy Vitamin D [25(OH)D] Levels, Supplemental Vitamin D, and Parathyroid Hormone Levels in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0419-11-FB
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Premature Infants
Keywords: vitamin D3; prematurity; parathyroid hormone; 25(OH)D; NICU hospitalization
MeSH Terms: conditions — Premature Birth | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 400 IU/day vitamin D (Active Comparator): Subjects will receive 400 IU/day of vitamin D3, as per current unit policy
  Interventions: Dietary Supplement: cholecalciferal
- 800 IU/day vitamin D3 (Experimental): Subjects will receive 800 IU/day vitamin D3
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferal — 400 IU/day
  Other Names: vitamin D3
  Arms: 400 IU/day vitamin D
Dietary Supplement: cholecalciferol — 800 IU/day D3
  Other Names: vitamin D3
  Arms: 800 IU/day vitamin D3

SUMMARY:
This study will determine levels of vitamin D supplementation to achieve goal serum 25-hydroxy vitamin D [25(OH)D] levels of 30 ng/mL, and to define serum 25(OH)D levels required to achieve suppression of parathyroid hormone in preterm newborn infants hospitalized in Newborn Intensive Care Nursery (NICU). Infants 23 weeks gestational age or greater will be randomized to two different levels of vitamin D supplementation: 400 IU vitamin D3/day, or 800 IU vitamin D3/day.

DETAILED DESCRIPTION:
The specific aims of this study are to determine levels of vitamin D supplementation to achieve goal serum 25(OH)D levels of 30 ng/mL, and to define serum 25(OH)D levels required to achieve suppression of parathyroid hormone in preterm newborn infants hospitalized in the Nebraska Medical Center Newborn Intensive Care Nursery (NICU). In this randomized, controlled trial, infants 23 weeks gestational age or greater will be randomized to two different levels of vitamin D supplementation: 400 IU vitamin D3/day, or 800 IU vitamin D3/day. As an exploratory aim, vitamin D binding protein levels (VDBP) will also be quantified in these infants.

ELIGIBILITY:
Inclusion Criteria:

* NICU hospitalized infants
* 23-32 weeks gestation

Exclusion Criteria:

* congential anomalies
* disorders of calcium metabolism
* inborn error of metabolism
* kidney disease
* liver disease
* use of steroids

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxy vitamin D [25(OH)D] Levels | 1 year
  Serum 25-hydroxy vitamin D [25(OH)D] levels will be compared between the two groups, vitamin D supplementation of 400 IU vitamin D3/day, or 800 IU vitamin D3/day. The specific aims of this study are to determine leves of vitamin D supplementation to achieve goal serum 25(OH)D levels of 30 ng/mL.

SECONDARY OUTCOMES:
Parathyroid Hormone Levels | 1 year
  Parathyroid hormone levels will be compared in between the two groups, vitamin D supplementation of 400 IU vitamin D3/day, or 800 IU vitamin D3/day.

CONTACTS AND LOCATIONS:
Overall Officials: Corrine K Hanson, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842